CLINICAL TRIAL: NCT06456372
Title: Digital Health Intervention for Children With ADHD: Improving Mental Health Intervention, Patient Experiences, and Outcomes
Brief Title: Digital Health Intervention for Children With ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Riverside (Other)
Collaborators: University of California, Irvine (Other); Chapman University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: R21HS028871/R33HS028871; R21HS028871 (NIH)
Record Dates: First submitted 2024-05-20; First posted 2024-06-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention)
- Digital Health Intervention Group (Experimental)
  Interventions: Behavioral: Digital Health Intervention Group

INTERVENTIONS:
Behavioral: Digital Health Intervention Group — Our digital health intervention (DHI) uses Patient-Centered Digital Healthcare Technologies (PC-DHT) to promote co-regulation (child/parent), capture patient data, support efficient healthcare delivery, enhance patient engagement, and facilitate shared decision-making, thereby improving access to timely and targeted mental health intervention for children at great risk for poor outcomes. This system will integrate treatment across multiple points of care and will enable health care providers and caregivers to share reliable and targeted information that will facilitate collaborative decision-making (e.g., making decisions about changing or titrating medications/dosages or shifting behavioral therapy and educational intervention targets) and improve patient experiences and outcomes.
  Arms: Digital Health Intervention Group

SUMMARY:
To conduct an RCT to evaluate the efficacy of the system, we will recruit 60 children (ages 8-12) with ADHD who will be randomized to either immediate (n=30) or delayed (n=30) treatment (i.e., a wait-list control group). Among those randomized to immediate treatment, half will be assigned to DHI (delivered via a smartwatch and smartphone application) and half will be assigned to an active control treatment as usual (TAU) group who will receive the smartwatch with no assigned activities, applications, or interventions on the devices. The intervention period will last 16 weeks; after a participant has been in the delayed treatment group for 16 weeks and has completed the post-waiting period assessment, he or she will be assigned to either the intervention or active control group. Thus, 30 participants will complete the intervention and 30 will complete the active control, with half of the total sample also completing a wait-list period.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5TR diagnosis of ADHD through prior medical or psychological evaluations at the time of admission to the program,
2. ability to complete questionnaires and use an app in English,
3. reported IQ of at least 80 in order to ensure that the participant has the cognitive skills needed to use the app, and
4. parent/guardian available to consent and provide feedback in English.

Exclusion Criteria:

* Failure to meet any of the inclusion criteria

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-02-22 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Child Self-Regulation - BASC-3 SRP, PRS, TRS | 1 Year
  Behavior Assessment System for Children - BASC-3 Self, Parent, and Teacher reports - The Behavior Assessment System for Children - Third Edition is an individually-administered, norm-referenced, comprehensive set of rating scales and forms designed to inform understanding of the behaviors and emotions of children and adolescents ages 2 years through 21 years, 11 months. Forms available in this system include Parent Rating Scales (PRS), Teacher Rating Scales (TRS), the Self-Report of Personality (SRP; 6 years through 21 years, 11 months), and the Parenting Relationship Questionnaire (PRQ).
  The TRS/PRS rater responds to items about observed behaviors by answering N for Never, S for Sometimes, O for Often, or A for Almost always. The SRP respondent answers items about personal thoughts and feelings experienced. SRP items have one of two response formats: T for True or F for False; or N for Never, S for Sometimes, O for Often, or A for Almost always.
ADHD Symptoms - BASC-3 SRP, PRS, TRS | 1 Year
  BASC-3 Self, Parent, and Teacher reports - The Behavior Assessment System for Children - Third Edition is an individually-administered, norm-referenced, comprehensive set of rating scales and forms designed to inform understanding of the behaviors and emotions of children and adolescents ages 2 years through 21 years, 11 months. Forms available in this system include Parent Rating Scales (PRS), Teacher Rating Scales (TRS), the Self-Report of Personality (SRP; 6 years through 21 years, 11 months), and the Parenting Relationship Questionnaire (PRQ). The TRS/PRS rater responds to items about observed behaviors by answering N for Never, S for Sometimes, O for Often, or A for Almost always. The SRP respondent answers items about personal thoughts and feelings experienced. SRP items have one of two response formats: T for True or F for False; or N for Never, S for Sometimes, O for Often, or A for Almost always.
ADHD Symptoms - Brown EF/A | 1 Year
  Brown Executive Function/Attention Scales (Parent and Self Reports) - The Brown Scales screen and assess impairments of executive functioning (EF) and attention. They assess a wide range of symptoms of EF impairments associated with ADHD/ADD. These normed rating scales elicit parent and teacher report for children ages 3-12 yrs. For 8-12 year olds, a normed self-report version is also available. The scales are organized into six clusters of EF (i.e., Activation, Focus, Effort, Emotion, Memory, Action) with items tapping severity not frequency. This measure contains context-specific items (e.g., difficulty remembering what has been read when assigned), includes DSM-5-TR ADHD symptoms, and aspects of EF impairments not in the disorder's diagnostic criteria. They are designed to be completed by various respondents who have knowledge about an individual's daily behaviors and who have had extended and frequent opportunities to observe the individuals' responses to environmental demands.
ADHD Symptoms - SWAN | 1 Year
  Strengths and Weakness of ADHD-symptoms & Normal-behavior Scale (SWAN: Self, Parent, and Teacher reports) - SWAN screens for ADHD in youth <18. It is completed by a parent/teacher & has 18 questions that compare a child's attention skills to others of the same age group, family, & school environment on skills like focusing attention, controlling anxiety, & inhibiting impulsive behavior during tasks that require prolonged mental effort & during daily activities. SWAN is based on observations of normal & abnormal attention skills in different populations & captures a range of behaviors. SWAN comprises 30 items measuring the full range of behavior, instead of only the pathological signs & symptoms of ADHD & measures behavioral characteristics representative of the attention skills of the general population. The seven-point response is scored from +3 to -3. Far below average = 3, below average = 2, slightly below average = 1; average = -1; above average = -2; & far above average = -3.
Parent Self-Regulation - BASC-3 PRQ | 1 Year
  BASC-3 Parenting Relationship Questionnaire (PRQ) - The BASC-3 PRQ is a measure of a parent's perspective on the parent's relationship with the child. It is standardized and normed and requires about 10-15 minutes for completion. It has 7 scales: Attachment, Communication, Discipline Practices, Involvement, Parenting Confidence, Satisfaction with School, Relational Frustration. Our primary focus will be on the Relational Frustration scale. Additional secondary analyses will be conducted to assess changes in parent behaviors. This scale can be administered remotely using Pearson's Q Global Remote Assessment Platform.
Engagement in Care - PAM Child | 1 Year
  The Patient Activation Measure® (PAM) is a 10- or 13-item survey that assesses an individual's knowledge, skills and confidence integral to managing one's own health and healthcare. PAM segments individuals into one of four activation levels, providing insight into health-related characteristics like attitudes, motivators and behaviors. Each item has four response options: "disagree strongly," "disagree," "agree" and "agree strongly." The PAM has a theoretical range from 0 to 100. Higher scores indicate greater activation.
Engagement in Care - PAM Parent | 1 Year
  Parent Patient Activation Measure (Parent PAM) - P-PAM was designed for use among caregivers of pediatric patients and requires parents to assess their knowledge, confidence, and willingness to act in regard to their child's health. The questionnaire aims to include a quantitative measure of all aspects of parent engagement on behalf of their child and also represents the individual level of engagement. Response options are on a four-point Likert scale ranging from (1) 'disagree strongly' to (4) 'agree strongly' or the option of (5) 'not applicable'. The total activation score was calculated on a continuous scale ranging from 0-100 and stratified into four levels of activation with higher scores corresponding to higher activation.
Perceptions of Shared-Decision Making and Treatment Collaborations - Child & Parent | 1 Year
  Working Alliance Inventory-Short Revised - The Working Alliance Inventory-Short Revised is a 12-item validated scale that evaluates the working relationship between a client and a clinician. A sample item reads, "I believe the way we are working with my problem is correct" and has a rating from 1 (seldom) to 5 (always).
Perceptions of Shared-Decision Making and Treatment Collaborations - Provider/Educator | 1 Year
  Working Alliance Inventory-Short Revised - The Working Alliance Inventory-Short Revised has a provider version of a 12-item validated scale that evaluates the working relationship between a client and a clinician. A sample item reads, "We are working on mutually agreed upon goals" and has a rating from 1 (seldom) to 5 (always). This scale has a version for other providers (e.g., physicians), which will be used for participants who are not providing mental health care to the child.

SECONDARY OUTCOMES:
Self-Efficacy - BASC-3 SRP | 1 Year
  BASC-3 Self-Report - The Behavior Assessment System for Children - The Behavior Assessment System for Children - Third Edition is an individually-administered, norm-referenced, comprehensive set of rating scales and forms designed to inform understanding of the behaviors and emotions of children and adolescents ages 2 years through 21 years, 11 months. Forms available in this system include Parent Rating Scales (PRS), Teacher Rating Scales (TRS), the Self-Report of Personality (SRP; 6 years through 21 years, 11 months), and the Parenting Relationship Questionnaire (PRQ).
  The TRS/PRS rater responds to items about observed behaviors by answering N for Never, S for Sometimes, O for Often, or A for Almost always. The SRP respondent answers items about personal thoughts and feelings experienced. SRP items have one of two response formats: T for True or F for False; or N for Never, S for Sometimes, O for Often, or A for Almost always.
Parent-Child Relationship - BASC-3 PRQ | 1 Year
  BASC-3 Parenting Relationship Questionnaire (PRQ) - The BASC-3 PRQ is a measure of a parent's perspective on the parent's relationship with the child. It is standardized and normed and requires about 10-15 minutes for completion. It has 7 scales: Attachment, Communication, Discipline Practices, Involvement, Parenting Confidence, Satisfaction with School, Relational Frustration. Our primary focus will be on the Relational Frustration scale. Additional secondary analyses will be conducted to assess changes in parent behaviors. This scale can be administered remotely using Pearson's Q Global Remote Assessment Platform.
Parent-Child Relationship - BASC-3 SRP | 1 Year
  BASC-3 Self Report (Relations with Parent scale) - The Behavior Assessment System for Children - Third Edition is an individually-administered, norm-referenced, comprehensive set of rating scales and forms designed to inform understanding of the behaviors and emotions of children and adolescents ages 2 years through 21 years, 11 months. Forms available in this system include Parent Rating Scales (PRS), Teacher Rating Scales (TRS), the Self-Report of Personality (SRP; 6 years through 21 years, 11 months), and the Parenting Relationship Questionnaire (PRQ).
  The TRS/PRS rater responds to items about observed behaviors by answering N for Never, S for Sometimes, O for Often, or A for Almost always. The SRP respondent answers items about personal thoughts and feelings experienced. SRP items have one of two response formats: T for True or F for False; or N for Never, S for Sometimes, O for Often, or A for Almost always.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Craig School, Irvine, California
  - UCR Psychiatry at Grindstaff Community School, Riverside, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cibrian, F., Cates, H., Guzman, K., Tavakoulnia, A., Shuck, S., Hayes, G., & Lakes, K.D. (2019). Should I wear a smartwatch? How children view wearables for behavior change. Workgroup on Interactive Systems in Healthcare, Chi'19.
- [Background] Cibrian, F. L., Lakes K.D., Schuck S, Tavakoulnia A, Guzman K, Hayes G. (2019). Balancing caregiver and child interactions to support the development of self-regulation skills using a smartwatch application. In Proceedings of the 2019 ACM International Joint Conference on Pervasive and Ubiquitous Computing and Proceedings of the 2019 ACM International Symposium on Wearable Computers (UbiComp/ISWC '19 Adjunct). ACM, New York, NY, USA, 459-460. https://doi.org/10.1145/3341162.3345612.
- [Background] Tavakoulnia A, Guzman K, Cibrian, F. L., Lakes K.D., Hayes G., Schuck S. (2019). Designing a wearable technology application for enhancing executive function skills in children with ADHD. In Proceedings of UbiComp/ISWC'19. ACM, New York, NY, USA. https://doi.org/10.1145/3341162.3343819
- [Background] Cibrian, F., Lakes, K.D., Tavakoulnia, A., Guzman, K., Schuck, S. & Hayes, G., (2020). Supporting self-regulation of children with ADHD using wearables: Tensions and design challenges. ACM CHI2020. https://doi.org/10.1145/3313831.3376837
- [Background] Cibrian, F., Doan, M., Jang, A., Khare, N., Chang, S., Li, A., Schuck, S., Lakes, K.D., & Hayes, G.R.].(2020). CoolCraig: A smart watch/phone application supporting co-regulation of children with ADHD. ACM CHI2020, 1-7. https://doi.org/10.1145/3334480.3382991
- [Background] Ankrah, E., Cibrian, F.L., Beltran, J.A., Tavakoulnia A., Silva L., Schuck S., Lakes, K. D., Hayes G. (2020). How children with ADHD understand health data from smartwatches. Proceedings of the 2020 CHI Conference on Human Factors in Computing Systems.
- [Background] Cibrian, F. L., Hayes, G., & Lakes, K.D. (2020). Research Advances in ADHD and Technology. USA: Morgan & Claypool Publishers.
- [Background] Silva, L.M., Cibrian, F., Bhattacharya, A., Ankrah, E., Monteiro, E., Beltran, J., Schuck, S.E.B., Epstein, D., Lakes, K.D., & Hayes, G.R. (2021). Adapting multi-device deployments during a pandemic: Lessons learned from two studies. IEEE Pervasive Computing.
- [Background] Cibrian FL, Monteiro E, Ankrah E, Beltran JA, Tavakoulnia A, Schuck SEB, Hayes GR, Lakes KD. Parents' perspectives on a smartwatch intervention for children with ADHD: Rapid deployment and feasibility evaluation of a pilot intervention to support distance learning during COVID-19. PLoS One. 2021 Oct 27;16(10):e0258959. doi: 10.1371/journal.pone.0258959. eCollection 2021. PMID 34705845
- [Background] Cibrian, F., Lakes, K.D., Schuck, S., & Hayes, G. (In Press). The potential impact of technologies supporting self-regulation in children with ADHD: A literature review. International Journal of Child-Computer Interaction.
- [Background] Lakes, K.D., Cibrian, F., Schuck, S., Nelson, M., & Hayes, G. (In Press). Digital health interventions for youth with ADHD: A mapping review. Computers in Human Behavior Reports.
- [Derived] Herrera N, Cibrian FL, Silva LM, Beltran JA, Schuck SEB, Hayes GR, Lakes KD. Digital health intervention for children with ADHD to improve mental health intervention, patient experiences, and outcomes: a study protocol. BMC Digit Health. 2024;2(1):78. doi: 10.1186/s44247-024-00134-4. Epub 2024 Nov 5. PMID 39507592